CLINICAL TRIAL: NCT05584605
Title: Changes in PERFusion and Cerebrovascular Reactivity Through Aerobic EXercise Training After Ischemic Stroke - a Proof of Concept Randomized Controlled Trial
Brief Title: Perfusion Augmentation Through Exercise
Acronym: PERFEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-00438
Record Dates: First submitted 2022-09-15; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Stroke, Ischemic
Keywords: cerebral perfusion; aerobic exercise
MeSH Terms: conditions — Ischemic Stroke | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic treadmill training (Experimental): Progressive graded, high-intensity aerobic treadmill training is delivered over 36 sessions at a frequency of 3x per week for 30-50 minutes of training per session over a period of 3 months. If possible, the training intensity is progressed from 40% to 80% of heart rate reserve, according to the supervising therapist.
  Interventions: Behavioral: Aerobic treadmill training
- stretching exercise (Active Comparator): The control intervention includes stretching exercise therapy similarly heart rate controlled within limits up to 20% of heart rate reserve over 36 sessions at a frequency of 3x per week for 30 minutes.
  Interventions: Behavioral: Stretching exercise

INTERVENTIONS:
Behavioral: Aerobic treadmill training — The intervention will be delivered based on the initial exercise testing and graded based by increasing the duration, speed and/or altitude of the treadmill training.
  Arms: aerobic treadmill training
Behavioral: Stretching exercise — Interventions, such as stretching, relaxation, passive soft-tissue technics (excl. manipulation) that do not elevate the heart rate above 20HRR
  Arms: stretching exercise

SUMMARY:
Large cerebral vessel occlusion is a common phenomenon in the general population and accounts for 13-35% of ischemic strokes. Chronic stenosis in the large cerebral arteries is associated with cerebral hypoperfusion, cognitive decline and an increased risk of stroke or recurrent stroke, respectively.

Even with upgrowth of surgical or endovascular interventions, mechanical reopening of the occluded vessels is often not possible. Alternative treatment opportunities include minimal-to-moderate blood pressure elevation (typically by ceasing antihypertensives) waiting for collateral circulation to develop spontaneously. Another conservative approach to increase cerebral perfusion is aerobic exercising. Physical activity has shown to lead to cerebral blood flow increase, especially in activated brain areas of healthy human and rat models. However, it is remains unknown, how physiological adaptation to physical activity expresses in persons after stroke due to large vessel occlusion. Herein, it is hypothesized that aerobic exercise facilitates the development of an extensive and functional vascular collateral network in persons with ischemic stroke and perfusion compromise.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients of 18 years of age or above
* Subjects after ischemic cerebral stroke (≥ 3 months) due to large vessel occlusion
* Subjects do not qualify for flow augmentation through ECIC bypass or endovascular treatment
* Persistent deficit in BOLD-CVR
* Functional Ambulatory Categories >2
* Discharged from hospitalization / inpatient rehabilitation
* Living independent before stroke (mRS ≤3)
* Written Informed Consent

Exclusion Criteria:

* Severe cardiac disease, such as instable angina pectoris, pericarditis, heart failure (New York Health Association > II°), or hemodynamically significant valvular dysfunction
* Complete arterial stenosis
* Peripheral artery disease with mild to moderate claudication at < 200m or 200-1000m of walking
* Contra-indication, such as a history of a seizure, prior electroconvulsive therapy, deep brain stimulators or other metal in the head, skull defect, pacemaker, neuroleptic medication
* Inability to follow the procedures of the study, e.g., due to language problems (unable to follow to stage commands), psychological disorders (major depression), and / or a neurodegenerative disease (dementia)
* Known or suspected non-compliance, documented drug, or alcohol abuse
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Brain imaging - cerebrovascular reactivity (CVR) by BOLD-fMRI | post-intervention (12 weeks)
  Functional brain tissue perfusion and tissue at risk based on cerebrovascular reactivity by blood oxygenation-level dependent functional magnetic resonance imaging (BOLD-fMRI), measured as the percentage BOLD signal change /mmHg CO2.

SECONDARY OUTCOMES:
Brain imaging - intravoxel incoherent motion (IVIM) | post-intervention (12 weeks)
  Functionality of brain microvasculature by measuring diffusion and perfusion components of tissue based on intravoxel incoherent motion
Brain imaging - NOVA-qMRI | post-intervention (12 weeks)
  Blood flow velocity based on non-invasive optimal vessel analysis quantitative magnetic resonance imaging
Brain imaging - Lesion volume | post-intervention (12 weeks)
  based on 3D T1 weighted imaging, 3D Fluid-Attenuated Inversion Recovery (FLAIR), Diffusion-Eighted Imaging (DWI)
Brain imaging - Collateral status | post-intervention (12 weeks)
  Collateral status based on 3D time of flight angiography (TOF)
Exercise stress testing | post-intervention (12 weeks)
  Cycle ergometer testing with spirometry
Six-Minute Walk Test (6MWT) | post-intervention (12 weeks) + follow-up (+3 months)
  Functional walking capacity in meters
Ten-Meter Walk Test (10MWT) | post-intervention (12 weeks) + follow-up (+3 months)
  Walking speed in m/s
Fugl-Meyer Assessment of the Lower Extremity (FMMA-LE) | post-intervention (12 weeks) + follow-up (+3 months)
  Stroke-specific motor impairment index to assess lower limb motor function with a total score ranging from 0 to 34 and higher scores indicating better performance.
Motricity Index of the Lower Extremity (MI-LE) | post-intervention (12 weeks) + follow-up (+3 months)
  Muscle strength assessment of three major muscle groups of the lower extremity with a total score ranging from 0 to 100 and higher scores indicating better performance.
5-Chair-Rise-Test | post-intervention (12 weeks) + follow-up (+3 months)
  Functional muscle strength, measured in seconds to complete the task.
International Physical Activity Questionnaire (IPAQ) | post-intervention (12 weeks) + follow-up (+3 months)
  self-reported physical activity
Montreal Cognitive Assessment (MoCA) | post-intervention (12 weeks) + follow-up (+3 months)
  Screening assessment of cognitive functions with a maximum score of 30 points.
Word list learning | post-intervention (12 weeks) + follow-up (+3 months)
  Assessment of memory function
Digit Span Test / Corsi block | post-intervention (12 weeks) + follow-up (+3 months)
  Assessment verbal and nonverbal working memory
Stroop test | post-intervention (12 weeks) + follow-up (+3 months)
  Assessment of executive function and inhibition
European Quality of Life 5 Dimensions 5 Level (5Q-5D-5L) | post-intervention (12 weeks) + follow-up (+3 months)
  Quality of life questionnaire that assesses 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) on a 5-level scale ranging from 1 - no, 2 - slight, 3 - moderate, 4 - severe to 5 - extreme problems or unstable to.

OTHER OUTCOMES:
Concomitant medications | post-intervention (12 weeks) + follow-up (+3 months)
  covariate

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Globas, MD, Principal Investigator — University Hospital and University of Zurich
Locations (3):
- Switzerland (3):
  - Ambulante Reha Triemli Zürich, Zurich
  - Klinik Lengg AG, Zurich
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No